CLINICAL TRIAL: NCT02460133
Title: Understanding HCV Reinfection Rates in an Incarcerated Population After Cure With Interferon Free HCV Treatment: A Pilot Project
Brief Title: Understanding HCV Reinfection Rates in an Incarcerated Population After Cure With Interferon Free HCV Treatment
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Provincial Correction Centre (PEI) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAIL-001
Record Dates: First submitted 2015-05-22; First posted 2015-06-02 (Estimated); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; Ritonavir; dasabuvir; ombitasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCV Genotype 1, with and without cirrhosis (Other)
  Interventions: Drug: Paritaprevir; Drug: Ritonavir; Drug: Dasabuvir; Drug: Ombitasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Paritaprevir
Drug: Ritonavir
Drug: Dasabuvir
Drug: Ombitasvir
Drug: Ribavirin — In genotype 1b individuals without cirrhosis, treatment will NOT include ribavirin.

SUMMARY:
This pilot study is crucial to determining whether treating individuals who are at high risk for transmission or re-infection will impact HCV reinfection rates. It will establish the feasibility of DAA treatment in corrections facilities, as well as delineate the underlying immune basis of HCV cure and reinfection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a blood-borne virus that causes both acute and chronic liver disease. Chronic HCV infection is associated with progressive liver disease and significant morbidity and mortality and represents a significant public health burden with approximately 150 million people infected worldwide. Until very recently, HCV treatment was extremely difficult for both clinicians and patients. Treatment strategies had debilitating side effects including dangerously low blood levels and clinical depression that often resulted in incomplete therapy and relatively infrequent cure (only 60-70% of individuals). In addition, the extended duration of therapy (up to one year) often precluded treatment for marginalized individuals with unstable life circumstances or intermittent incarceration.

Within the last 4 years, new direct acting antivirals (DAA) have been licensed for the treatment of HCV infection. These newly approved regimens are short (12 weeks), extremely safe, well tolerated and result in cure rates in excess of 90%.

HCV cure is defined as undetectable serum HCV viral load 12 weeks after finishing therapy. This is also termed 12 week sustained virologic response or SVR12.

In Canada, over 240,000 individuals have HCV, and the majority of new HCV infections occur through intravenous drug use. Many of these individuals encounter the federal and/or provincial corrections system at some point in their lifetime, and it is estimated that up to 80% of injection drug users (IVDU) practice needle sharing. Incarcerated individuals are a vulnerable, high risk population who are generally excluded from clinical studies and access to novel classes of antiviral therapies.

If all individuals were diagnosed, treated and cured, incident and chronic HCV infection within the incarcerated population would likely be greatly reduced (a type of harm reduction or treat to prevent strategy). Additionally, there may be an immunologic rationale for reduced rates of reinfection after viral cure with these therapies, and immune investigations in this study address this issue. Essentially, this study asks whether treatment of the majority of HCV positive individuals in a discrete population is harm reduction in and of itself. That is, individuals may have decreased susceptibility to HCV infection because of increased immunity and the population may see decreased reinfection rates because of reduced viral reservoir in the local community.

This novel pilot study is crucial to determine whether treating individuals who are at high risk for transmission or re-infection will impact HCV reinfection rates. This study will establish the feasibility of DAA treatment in corrections facilities, as well as delineate the underlying immune basis of HCV cure and reinfection.

ELIGIBILITY:
Inclusion Criteria:

* An offender at the PEI Provincial Correction Centre during the enrollment time
* Male, 18 -70 years of age, inclusive, at time of screening
* Chronic HCV genotype 1 infection
* HCV infection, as demonstrated by positive HCV immunosorbant assay and detectable HCV viral load
* No evidence of decompensated liver disease (refractory ascites, variceal bleed within 1 year, active hepatic encephalopathy or Child-Pugh score greater than 6)
* HIV negative
* Males must be abstinent from sexual intercourse, surgically sterile or agree to practice two effective forms of birth control from those listed below, throughout the course of the study, starting with Study Day 1 and for 7 months after the last dose of study drug (or per local RBV label):

  * Partner(s) using an IUD (intrauterine device),
  * Partner(s) using oral, injected, or implanted methods of hormonal contraceptives,
  * Subject and/or partner(s) using condoms, contraceptive sponge, or diaphragm with spermicidal jellies or creams.
* Subjects must be able to understand and adhere to the study visit schedule and all other protocol requirements
* Must voluntarily sign and date an informed consent form, approved by a Research Ethics Board prior to the initiation of any screening or study specific procedures

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any drug
* Positive test result at screening for Hepatitis B surface antigen
* Prior therapy with direct acting antivirals for the treatment of HCV
* Evidence of decompensated liver disease (current or past refractory ascites, variceal bleed within 1 year, active hepatic encephalopathy)
* HIV positive screening test
* Unwilling to follow up for 48 weeks after treatment completion
* Use of any herbal supplements (including milk thistle) within 2 weeks or 10 half-lives of the respective supplement, whichever is longer, prior to the first dose of study drug
* HCV genotype performed during screening indicating unable to genotype or co-infection with any other HCV genotype
* Use of any medications contraindicated for use with the study regimen
* Clinically significant abnormalities, other than HCV-infection, based upon the results of a medical history, physical examination, vital signs, and laboratory profile that make the subject an unsuitable candidate for this study in the opinion of the investigator
* Serum Alpha-Fetoprotein (AFP) > 200 ng/mL at screening
* Any cause of liver disease other than chronic HCV-infection, including but not limited to the following:

  * Hemochromatosis
  * Alpha-1 antitrypsin deficiency
  * Wilson's disease
  * Autoimmune hepatitis
  * Alcoholic liver disease
  * Nonalcoholic steatohepatitis
  * Drug-related liver disease
* Screening laboratory analyses showing any of the following abnormal laboratory results:

  * ALT > 5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) > 5 × ULN
  * Calculated creatinine clearance (using Cockcroft-Gault method) < 60 mL/min
  * Albumin 25 g/L
  * Prothrombin time/International normalized ratio (INR) > 2.3.
  * Hemoglobin < LLN
  * Platelets < 60,000 cells per mm3
  * Absolute neutrophil count (ANC) < 1500 cells/μL
  * Total bilirubin ≥ 51 umol/L
* History of solid organ transplantation.
* Receipt of any investigational product within a time period equal to 10 half-lives of the product, if known, or a minimum of 6 weeks prior to study drug administration.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive paritaprevir, dasabuvir, ombitasvir, ritonavir and/or RBV.
* Current enrollment in another clinical study, prior enrollment in this study, or previous exposure to paritaprevir, ombitasvir, or dasabuvir. Concurrent participation in a non-interventional, epidemiologic or registry trials may be permitted with approval of the principal investigator.
* The use of colony stimulating factors, such as granulocyte colony stimulating factor (GCSF) or erythropoietin within 2 months of the screening period.
* Uncontrolled clinically significant cardiac, respiratory (except mild asthma), hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness, which is unrelated to the hepatic disease.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Re-infection rate in individuals treated with DAA therapy | 1 year following treatment.
  This will require HCV quasispecies determination at baseline and in potentially re-infected individuals. Re-infection will require demonstration of HCV RNA above level of detection after SVR12 with a phyogenetically distinct HCV species.

SECONDARY OUTCOMES:
Percentage of subjects with sustained virologic response at 12 weeks post treatment | 12 Weeks post treatment
Change in fibrosis measured by transient elastography | From day 0 to the end of follow-up
Global and HCV-specific T cell function before and after treatment with DAA therapy. | From day 0 to end of follow-up
Global and HCV-specific B cell function before and after treatment with DAA therapy. | From day 0 to end of follow-up
Global and HCV-specific NK cell function before and after treatment with DAA therapy. | From day 0 to end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Barrett, MD PhD FRCPC, Principal Investigator — Department of Medicine, Division of Infectious Diseases, Nova Scotia Health Authority, Dalhousie University